CLINICAL TRIAL: NCT03024749
Title: Surgical Intervention of Spinal Arteriovenous Malformations and Fistulas: Multicenter Prospective Cohort Study
Brief Title: Surgical Intervention of Spinal Arteriovenous Malformations and Fistulas
Acronym: SUIT-SAVM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hongqi Zhang, MD (Other)
Collaborators: Beijing Tiantan Hospital (Other); Beijing Tsinghua Chang Gung Hospital (Other); Tianjin Medical University General Hospital (Other); Peking University Third Hospital (Other); Chinese PLA General Hospital (Other); Beijing Hospital (Other Government); General Hospital of Chinese Armed Police Forces (Other); Beijing Haidian Hospital (Other); China Rehabilitation Research Center (Other Government)
Responsible Party: Sponsor-Investigator, Hongqi Zhang, MD, Director of Neurosurgery, Xuanwu Hospital, Beijing
Organization: Xuanwu Hospital, Beijing (Other)
Other Study IDs: D161100003816001
Record Dates: First submitted 2016-12-27; First posted 2017-01-19 (Estimated); Last update posted 2017-06-06 (Actual); Status verified 2017-06

CONDITIONS: Spinal Cord Vascular Diseases
Keywords: Spinal Arteriovenous Malformation; Spinal Arteriovenous Fistula
MeSH Terms: conditions — Spinal Cord Vascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Spinal arteriovenous fistulas (AVFs) and arteriovenous malformations (AVMs) are complex neurosurgical lesions that are very challenging to manage. Spinal vascular malformations account for 3%-4% of all intradural spinal cord mass lesions. Over the last few decades our understanding of these lesions has dramatically increased thanks to neuroimaging technology (e.g. spinal angiography and indocyanine green angiography). Various treatment modalities including conservative observation, endovascular embolization, microsurgical resection, radiation therapy, and combined therapies have been reported. The treatment for these AVMs and AVFs depends on their location, the type of malformation, the area of the spine involved, and the condition of the patient at the time of treatment. Due to the rarity of these spinal vascular lesions, reports of their management and outcomes have been limited to small series and case reports. And the rates of obliteration and outcomes are not satisfactory, especially the spinal AVMs. Spinal vascular lesions are rare but represent a formidable challenge for the treating neurosurgeon.The purpose of this study is to establish multimodality treatment mode and evaluate the anatomical cure rate and functional preservation rate.

DETAILED DESCRIPTION:
This is a multicenter, prospective, observational, registration study. There are nine centers involved in the study. The investigators set up a more detailed classification system for spinal vascular malformations. In accordance with inclusion criteria and exclusion criteria, this cohort study will include 380 samples in the study period of three years. According to the spinal angiography, the correct diagnosis and treatment strategy will be made. The minimally invasive surgical treatment methods and new techniques will be adopted such as spinal superselective angiography, preoperative embolization, intraoperative electrophysiological monitoring, intraoperative angiography, etc. All the enrolled patients will be visited a total of four times, postoperative day 1 and postoperative day 7, followed up postoperative 3 months and 12 months. The anatomical cure rate and spinal cord function will be assessed objectively. All data will be recorded in the network database platform.

ELIGIBILITY:
Inclusion Criteria:

* patient diagnosed with spinal vascular diseases including

  * intradural arteriovenous malformation,
  * intradural arteriovenous fistula,
  * dural arteriovenous fistula,
  * extradural arteriovenous malformation,
  * paravertebral arteriovenous malformation,
  * paravertebral arteriovenous fistula,
  * cobbs' syndrome,
  * other spinal arteriovenous metameric syndromes involve the spinal cord.
* patient not received surgical or interventional treatment before
* patient with normal cardiac, renal and hepatic function
* patient capable of understanding the content of the patient information / Informed Consent Form
* patient willing and able to participate in the registry

Exclusion Criteria:

* patient received surgical treatment or interventional treatment before
* patient is pregnant
* patient allergic to iodine
* patient unable to complete follow-up
* patient with cerebral lesions
* patient with other spinal lesions
* patient with cardiac, renal or hepatic dysfunction

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with spinal AVMs/AVFs
Sampling Method: Non-Probability Sample
Enrollment: 380 (Estimated)
Dates: Start 2016-12-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of the spinal cord function | 1 day before operation and 12 months postoperative
  American Spinal Injury Association(ASIA) Score for evaluating the spinal cord function.Indexes (ASIA score) at baseline (1 day before operation) and 12 months follow-up will be collected, then the change from preoperative to 12 months follow-up will be assessed.

SECONDARY OUTCOMES:
Anatomic obliteration rate | 3 months post operation
  the anatomic obliteration rate is determined by angiography 3 months post operation.
American Spinal Injury Association(ASIA) Score | 1 week, 3 months, 6 months, 12 months post operation
Modified Aminoff & Logue's Scale (mALS) | 1 week, 3 months, 6 months, 12 months post operation
Modified Denis Pain and Numbness Scale (mDPNS) | 1 week, 3 months, 6 months, 12 months post operation
Incidence of perioperative complications | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Zhang Hongqi, MD, Study Director — Neurosurgical Department, Xuanwu Hospital, Beijing
Locations (1):
- Tao Hong, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lee YJ, Terbrugge KG, Saliou G, Krings T. Clinical features and outcomes of spinal cord arteriovenous malformations: comparison between nidus and fistulous types. Stroke. 2014 Sep;45(9):2606-12. doi: 10.1161/STROKEAHA.114.006087. Epub 2014 Jul 15. PMID 25028446
- [Background] Rangel-Castilla L, Russin JJ, Zaidi HA, Martinez-Del-Campo E, Park MS, Albuquerque FC, McDougall CG, Nakaji P, Spetzler RF. Contemporary management of spinal AVFs and AVMs: lessons learned from 110 cases. Neurosurg Focus. 2014 Sep;37(3):E14. doi: 10.3171/2014.7.FOCUS14236. PMID 25175433
- [Background] Gross BA, Du R. Spinal glomus (type II) arteriovenous malformations: a pooled analysis of hemorrhage risk and results of intervention. Neurosurgery. 2013 Jan;72(1):25-32; discussion 32. doi: 10.1227/NEU.0b013e318276b5d3. PMID 23096418
- [Background] Gross BA, Du R. Spinal pial (type IV) arteriovenous fistulae: a systematic pooled analysis of demographics, hemorrhage risk, and treatment results. Neurosurgery. 2013 Jul;73(1):141-51; discussion 151. doi: 10.1227/01.neu.0000429848.91707.73. PMID 23615108